CLINICAL TRIAL: NCT01435434
Title: Mononucleotide Autologous Stem Cells and Demineralized Bone Matrix in the Treatment of Non Union/Delayed Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: lieb001-CTIL-HMO
Record Dates: First submitted 2011-09-04; First posted 2011-09-16 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Non Union/Delayed Fractures
Keywords: subjects sustaining Non union/delayed fractures and requiring surgical intervention for treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sepax, ignite, fracture healing (Experimental): the mesenchymal cells will be separated by sepax separation system and demineralized bone matrix will be done using IGNITE INJECTABLE REPAIR GRAFT
  Interventions: Device: the Sepax is a tool to standardize adult stem cell. Ignite ®ICS injectable scaffold manufactured by Wright Medical Technology.

INTERVENTIONS:
Device: the Sepax is a tool to standardize adult stem cell. Ignite ®ICS injectable scaffold manufactured by Wright Medical Technology.

SUMMARY:
The study is a prospective, trial to test the safety and feasibility of injecting autologous, isolated, sterile centrifuged NBMC, and Ignite® DBM in the treatment of high risk non union/delayed fractures. Another objective is to turn this procedure to a standard care protocol in our department .

ELIGIBILITY:
Inclusion Criteria:

1. Ages: 18 to 65
2. Males- not involved in active military duty.
3. Females-non child bearing potential, or females of child-bearing potential who have a negative pregnancy test (hCG urine) within 72 hours of informed consent.
4. Subjects must be available for follow-up for 1 year. 5"Hard to heal" fracture include the following: A. Fracture of the distal third of the tibial bone B. Segmental or open (II, IIIa an IIIB) fractures of the the tibia or femur diaphysis C.Articular fracture of the lower extremity (distal femur, tibial plateau and tibial pilon fractures) with significant metaphyseal comminution and/or bone loss.

Exclusion Criteria:

1. Active systemic or local infection.
2. History of malignancy, radiotherapy, or chemotherapy for malignancy (except BCC of the skin)
3. Pathological Fractures.
4. Prior Fracture or Prior operation in the current fracture

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
clinical and radiological bony union at 3 months and 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Jerusalem, Israel